CLINICAL TRIAL: NCT05947461
Title: Rectal Disclofenac Versus Indomethacin for Prevention of Post-ERCP Pancreatitis (DIPPP): a Multicentre, Double-blind, Randomised, Controlled Trial
Brief Title: Prevention of Post-ERCP Pancreatitis by Indomethacin Vs Diclofenac
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The data from the interim analysis showed a opposite trend predicting possible of benefit of indomethacin and conditional power analysis revealed a low probability of confirming the benefit of diclofenac if this trial will be continued.
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20232165-C-1
Record Dates: First submitted 2023-06-20; First posted 2023-07-17 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-07

CONDITIONS: Post-ERCP Acute Pancreatitis; NSAIDs; Indomethacin; Diclofenac; Endoscopic Retrograde Cholangiopancreatography
MeSH Terms: interventions — Diclofenac; Indomethacin

STUDY DESIGN:
Intervention Model Description: Participants in the interventional group received 100mg rectal dicfenac
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- diclofenac group (Experimental): Patients without contraindications in diclofenac group received 100mg rectal diclofenac 30 mins before ERCP procedure.
  Interventions: Drug: 100mg diclofenac
- Indomethacin group (Active Comparator): Patients without contraindications in indomethacin group received 100mg rectal indomethacin 30 mins before ERCP procedure.
  Interventions: Drug: 100mg indomethacin

INTERVENTIONS:
Drug: 100mg diclofenac — All patients without contraindications should receive 100mg rectal diclofenac 30mins before ERCP procedure
  Arms: diclofenac group
Drug: 100mg indomethacin — All patients without contraindications should receive 100mg rectal indomethacin 30mins before ERCP procedure
  Arms: Indomethacin group

SUMMARY:
Post-ERCP pancreatitis (PEP) is the most common complication after ERCP, which was associated with occasional mortality, prolonged hospital days and increased health costs. Some studies investigated the effectiveness of different Nonsteroidal antiinflammatory drugs (NSAIDs) for prevent PEP. However, several high-quality RCTs and meta-analyses consistently demonstrated only100mg rectal indomethacin or diclofenac significantly reduced PEP incidence compared with placebos. Thus, European Society of Gastrointestinal Endoscopy, American Society for Gastrointestinal Endoscopy and Japanese Society of Hepato-Biliary-Pancreatic surgery guidelines recommended rountine administration of 100mg rectal indomethacin or diclofenac in unselected patients who underwent ERCP.

Up to date, the mechanisms of NSAIDs in preventing pancreatitis were not fully elucidated. Diclofenac and Indomethacin showed similar inhibitory effects in phospholipase A2 and cyclooxygenase pathways. And the peak concentration of diclofenac and indomethacin both occurs between 30 and 90 min after rectal administration. However, diclofenac may be a stronger inhibitor of other pancreatitis-related imflammatory siginals (e.g. nuclear factor kappa-B) than indomethacin. Recently, several meta-analyses found 100mg rectal diclofenac to be more efficacious than 100mg rectal indomethacin. Despite these data, there is no conclusive evidence to prove that rectal diclofenac could provide incremental benefits over indomethacin from high-quality randomized, controlled trials. Therefore, the investigators conducted a multicenter, double-blind, randomized, controlled clinical trial to evaluate the efficacy of rectal diclofenac versus indomethacin for the prevention of post-ERCP pancreatitis in average-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-90 years old patients planned to undergo ERCP

Exclusion Criteria:

* Allergy to NSAIDs
* The administration of NSAIDs within 7 days
* Not suitable for NSAIDs administration (gastrointestinal hemorrhage within 4 weeks, renal dysfunction [Cr >1.4mg/dl=120umol/l]; presence of coagulopathy before the procedure)
* Previous biliary sphincterotomy and papillary large balloon dilation
* Acute pancreatitis within 3 days before ERCP
* Hemodynamical instability
* Pregnancy or lactation
* Unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1204 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-22 (Actual); Study Completion 2024-06-22 (Actual)

PRIMARY OUTCOMES:
Rate of post-ERCP Pancreatitis | 30 days
  The diagnosis of post-ERCP pancreatitis was confirmed if there was new onset of upper abdominal pain associated with an increased amylase or lipase level of at least 3 times the upper limit of normal range at 24 hours after ERCP, accompanied with extension of hospitalization for at least 2 nights.

SECONDARY OUTCOMES:
Rate of moderate or severe PEP | 30 days
  The severity classification of post-ERCP pancreatitis was defined according to the Cotton Criteria. Mild PEP: with an extension of hospitalization period of 2-3 days; Moderate PEP: with an extension of hospitalization period of 4-10 days; Severe PEP: with an extension of more than 10 days, or hemorrhagic pancreatitis, phlegmon, or pseudocyst, intervention (percutaneous drainage or surgery), or death.
Rate of Overall ERCP-related complications | 30 days
  ERCP-related complications include post-ERCP pancreatitis, gastrointestinal bleeding, perforation or infection according to Cotton Criteria.
Rate of patients with different severity of pancreatitis evaluated by revised Atlanta criteria | 30 days
Rate of NSAIDs-related complications | 30 days
  NSAIDs-related complications include: acute kidney injury, allergic reaction, gastrointestinal bleeding, myocardial infarction, cerebrovascular accident, and death

OTHER OUTCOMES:
Rate of ERCP-related perforation | 30 days
  Perforation was established according to Cotton criteria
Rate of ERCP-related infection | 30 days
  Infection was established according to Cotton criteria
Rate of ERCP-related bleeding | 30 days
  Bleeding was established according to Cotton criteria
Rate of mortality | 30 days
Number of hospital days after ERCP | 180 days

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Department of gastroenterology, Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Department of Gastroenterology, Fujian Medical University Xiamen Humanity Hospital, Xiamen, Fujian
  - Department of Gastroenterology, The 980th Hospital of the PLA Joint Logistics Support Force, Shijiazhuang, Hebei
  - Department of Gastroenterology, Huaihe Hospital of Henan University, Kaifeng, Henan
  - Department of Hepatobiliary Surgery, General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Department of Gastroenterology,The 986th Hospital of Xijing Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Air Force Military Medical University, China, Xi'an, Shaanxi
  - Deparment of hepatobiliary surgery, The First Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Department of Gastroenterology and Endoscopy, Department of Gastroenterology and EndoscopyThe Third Affiliated Hospital of Naval Military Medical University, Shanghai, Shanghai Municipality
  - Department of Gastroenterology, General Hospital of Xinjiang Military Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Kang X, Guo X, Chen Z, Zhou Z, Luo H, Lu Y, Lou L, Guo X, Pan Y. The Incidence and Severity of Post-ERCP Pancreatitis in Patients Receiving Standard Administration of NSAIDs: a Systematic Review and Meta-analysis. J Gastrointest Surg. 2022 Nov;26(11):2380-2389. doi: 10.1007/s11605-022-05399-6. Epub 2022 Aug 8. PMID 35941494
- [Background] Akshintala VS, Sperna Weiland CJ, Bhullar FA, Kamal A, Kanthasamy K, Kuo A, Tomasetti C, Gurakar M, Drenth JPH, Yadav D, Elmunzer BJ, Reddy DN, Goenka MK, Kochhar R, Kalloo AN, Khashab MA, van Geenen EJM, Singh VK. Non-steroidal anti-inflammatory drugs, intravenous fluids, pancreatic stents, or their combinations for the prevention of post-endoscopic retrograde cholangiopancreatography pancreatitis: a systematic review and network meta-analysis. Lancet Gastroenterol Hepatol. 2021 Sep;6(9):733-742. doi: 10.1016/S2468-1253(21)00170-9. Epub 2021 Jun 30. PMID 34214449
- [Background] Luo H, Zhao L, Leung J, Zhang R, Liu Z, Wang X, Wang B, Nie Z, Lei T, Li X, Zhou W, Zhang L, Wang Q, Li M, Zhou Y, Liu Q, Sun H, Wang Z, Liang S, Guo X, Tao Q, Wu K, Pan Y, Guo X, Fan D. Routine pre-procedural rectal indometacin versus selective post-procedural rectal indometacin to prevent pancreatitis in patients undergoing endoscopic retrograde cholangiopancreatography: a multicentre, single-blinded, randomised controlled trial. Lancet. 2016 Jun 4;387(10035):2293-2301. doi: 10.1016/S0140-6736(16)30310-5. Epub 2016 Apr 28. PMID 27133971
- [Derived] Kang X, Xia M, Wang J, Wang X, Luo H, Qin W, Liang Z, Zhao G, Yang L, Sun H, Tao J, Ning B, Zhong L, Zhang R, Ma X, Zhao J, Yue L, Jin H, Kang C, Ren G, Liang S, Wang H, Wang L, Nie Y, Wu K, Fan DM, Pan Y. Rectal diclofenac versus indomethacin for prevention of post-ERCP pancreatitis (DIPPP): a multicentre, double-blind, randomised, controlled trial. Gut. 2025 Jun 6;74(7):1094-1102. doi: 10.1136/gutjnl-2024-334466. PMID 40113243